CLINICAL TRIAL: NCT06127342
Title: Exercise and Emotional Learning in Posttraumatic Stress Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christal L Badour (Other)
Collaborators: University of Texas at Austin (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Christal L Badour, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90369; R61MH132722 (NIH)
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: PTSD
Keywords: Interpersonal Violence; Exercise
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moderate Intensity Exercise (Experimental): Visit 1: Participants will complete study screening, PTSD assessments, and provide written narrative for a traumatic event and a neutral control event.
  Visit 2: Participants will complete baseline structural MRI scans before completing 8 trials of imaginal exposure - 4 neutral then 4 trauma narratives - with psychophysiological and fMRI measurement. Following completion of the imaginal exposure task, the participant will perform Moderate-Intensity Exercise (30-min at 70-75% max HR with 5-min warm-up and 5-min cool-down at 40-50% max HR), on a stationary bike.
  Visit 3: Participants will complete the same imaginal exposure with measurement of psychophysiology, fMRI, and subjective emotional responding.
  Interventions: Behavioral: Moderate Intensity Exercise
- Low Intensity Exercise (Active Comparator): Visit 1: Participants will complete study screening, PTSD assessments, and provide written narrative for a traumatic event and a neutral control event.
  Visit 2: Participants will complete baseline structural MRI scans before completing 8 trials of imaginal exposure - 4 neutral then 4 trauma narratives - with psychophysiological and fMRI measurement. Following completion of the imaginal exposure task, the participant will perform Low-Intensity Exercise (control; 40-mins at 40-50% max HR),on a stationary bike.
  Visit 3: Participants will complete the same imaginal exposure with measurement of psychophysiology, fMRI, and subjective emotional responding.
  Interventions: Behavioral: Low Intensity Exercise

INTERVENTIONS:
Behavioral: Moderate Intensity Exercise — Participants will wear a heartrate monitor and cycle on a stationary bike at a slow speed for 5 minutes, then slowly cycle on a stationary bike for 30 minutes, then cycle on the stationary bike at a slow speed for 5 minutes.
  Arms: Moderate Intensity Exercise
Behavioral: Low Intensity Exercise — Participants will wear a heartrate monitor and cycle on a stationary bike at a slow speed for 40 minutes.
  Arms: Low Intensity Exercise

SUMMARY:
The goal of this clinical trial is to test how exercise affects learning and memory processes relevant to the treatment of PTSD. Participants will complete a baseline intake followed by two experimental sessions. During the first experimental session, participants will undergo an MRI session of imaginal exposure to traumatic memory cues followed by 30-minutes of moderate intensity exercise or low intensity exercise. Participants will complete a second session of imaginal exposure with MRI 24 hours later.

DETAILED DESCRIPTION:
The proposed project would build on our published pilot data and animal models to demonstrate that moderate intensity physical exercise delivered after exposure therapy engages fear circuitry and enhances the consolidation of therapeutic safety learning, thereby enabling enhanced symptom reduction for PTSD. Adults with PTSD related to interpersonal violence (IPV) exposure would complete an initial session of imaginal exposure to traumatic memory cues adapted for an MRI setting. This would be followed by 30-mins of moderate intensity exercise or low intensity exercise control. Participants would return 24-hrs later to complete a second session of imaginal exposure with MRI.

ELIGIBILITY:
Inclusion Criteria:

* Adults with PTSD related to interpersonal violence

Exclusion Criteria:

* Active or recent (within the last 3 months) severe substance use disorder(s)
* Active or recent (within the last 3 months) suicidal, psychotic, or manic symptoms/ episodes
* Significant developmental disabilities
* Current daily benzodiazepine or stimulant use with inability to abstain for study sessions
* Recent changes in psychiatric medication or trauma focused cognitive-behavioral therapy (CBT) (past 4-weeks)
* Medical condition(s) that prohibit exercise
* History of traumatic brain injury (TBI) with loss of consciousness > 30 mins
* Magnetic resonance imaging (MRI) contraindication(s)
* Positive pregnancy test
* History of seizure disorder
* Spontaneous seizure(s) within the last 3 months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in participant subjective emotional ratings | 24 hours
  Participant anxiety will be measured at baseline and after each imagery trial using a 10-point Likert-type scale with higher scores indicative of more subjective anxiety.
Change in Heart Rate | 24 hours
  Participant heart rate will be measured at baseline and after each imagery trial using a Biopac MP160 system
Change in Fear Circuit Blood Oxygen Level-Dependent (BOLD) Response | 48 hours
  Blood Oxygen Level-Dependent (BOLD) imaging will be measured during each imagery trial

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Adams, Jr., PhD, Principal Investigator — University of Kentucky; Christal Badour, PhD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - University of Texas, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Demographic, clinical, psychophysiological, and MRI data will be acquired from adults with PTSD related to interpersonal violence (IPV). All data will be de-identified prior to receipt by the repository, but the information needed to generate a global unique identifier for the National Institute of Mental Health (NIMH) Data Archive (NDA) will be collected for each subject. Sufficient data from this project will be preserved to enable sharing via NDA data of sufficient quality to validate and replicate research findings described in the Aims. NIMH requires data measured from human subjects to be shared using the NDA.
Supporting Information: Analytic Code